CLINICAL TRIAL: NCT01575795
Title: Standard (180mg) Versus Double (360mg) Loading Dose of Ticagrelor in Patients With ST-elevation Myocardial Infarction (STEMI), Undergoing Primary Percutaneous Coronary Intervention (PCI): a Multi-center Randomized Parallel Pharmacodynamic Study.
Brief Title: Standard (180mg) Versus Double (360mg) Loading Dose of Ticagrelor in Patients With ST-elevation Myocardial Infarction (STEMI), Undergoing Primary Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-10
Record Dates: First submitted 2012-04-09; First posted 2012-04-11 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: Ticagrelor; ST elevation acute myocardial infarction; Platelet reactivity
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor 180mg loading dose (Active Comparator): Ticagrelor 180mg loading dose
  Interventions: Drug: Ticagrelor
- Ticagrelor 360mg loading dose (Experimental): Ticagrelor 360mg loading dose
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor 360mg loading dose immediately pre prior percutaneous coronary intervention 360mg loading dose
  Arms: Ticagrelor 360mg loading dose
Drug: Ticagrelor — Ticagrelor 180mg loading dose 180mg loading dose
  Arms: Ticagrelor 180mg loading dose

SUMMARY:
This is a multi-center, prospective, randomized, single-blind, investigator initiated, pharmacodynamic study of parallel design, performed at 3 institutions (Patras University Hospital; Evangelismos Athens General Hospital; Gennimatas Athens General Hospital).

Patients with ST elevation myocardial infarction (symptom onset < 12 hours), undergoing primary percutaneous coronary intervention, who are antiplatelet naïve (Group A) or present high residual PR (defined as PRU ≥ 208) immediately before primary percutaneous coronary intervention, will be randomized after informed consent, in a 1:1 ratio to either:

Ticagrelor 180mg loading dose (LD), followed by a 90mg x2 maintenance dose (MD )starting 12±6 hours post LD Or Ticagrelor 360mg loading dose (LD), followed by a 90mg x2 maintenance dose (MD) starting 12±6 hours post LD Platelet reactivity assessment will be performed at randomization (Hour 0) and at 0.5, 1, 2, 4 hours after randomization, using the VerifyNow assay, in platelet reactivity units (PRU).

Documentation of major adverse cardiac events (death, myocardial infarction, stroke, urgent revascularization procedure with PCI or CABG) and bleeding (according to Bleeding Academic Research Consortium criteria) will be performed until patient's discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Patients with STEMI (onset of pain < 12 hours) with indication for primary PCI
3. Antiplatelet naïve or presenting HTPR (≥ 208 PRU) immediately before primary percutaneous coronary intervention
4. Informed consent obtained in writing

Exclusion Criteria

* Pregnancy
* Breastfeeding
* Inability to give informed consent or high likelihood of being unavailable until the Day 5
* Cardiogenic shock
* Major periprocedural complications (death, stent thrombosis, vessel perforation, arrhythmias requiring cardioversion, temporary pacemaker insertion or intravenous antiarrhythmic agents, respiratory failure requiring intubation, vascular injury (arteriovenous shunt, retroperitoneal bleeding), major bleeding (need for bood transfusion or drop in haemoglobin post-PCI by ≥ 5 gr/ dl or intracranial bleeding).
* Unsuccessful PCI (residual stenosis > 30% or flow < ΤΙΜΙ 3)
* Known hypersensitivity to ticagrelor
* History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 3 months.
* Other bleeding diathesis, or considered by investigator to be at high risk for bleeding
* Any previous history of stroke, intracranial hemorrhage or disease (neoplasm, arteriovenous malformation, aneurysm).
* Thrombocytopenia (< 100.000/μL) at randomization
* Anaemia (Hct < 30%) at randomization
* Polycytaemia (Hct > 52%) at randomization
* Periprocedural IIb/IIIa inhibitors administration
* Thrombolysis administration
* Recent (< 6 weeks) major surgery or trauma, including GABG.
* Subjects receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors that cannot be discontinued for the duration of the study.
* Concomitant oral or IV therapy with strong CY P3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazana vir, grapefruit juice N1 L/d), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or strong CYP3A inducers (rifampin/rifampicin, phenytoin, carbamazepine).
* Increased risk of bradycardiac events.
* Dialysis required.
* Severe uncontrolled chronic obstructive pulmonary disease
* Known severe hepatic impairment

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
platelet reactivity at 1 hour post randomization in Group A, between the 2 treatment arms. | 1 hour
  platelet reactivity at 1 hour post randomization in Group A, between the 2 treatment arms.

SECONDARY OUTCOMES:
1. Platelet reactivity at 1 hour post randomization in Group B, between the 2 treatment arms. | 1 hour
  1. Platelet reactivity at 1 hour post randomization in Group B, between the 2 treatment arms.
2. Platelet reactivity at 0.5 hour post randomization between the 2 treatment arms separately for Group A and B | 0.5 hour
  Platelet reactivity at 0.5 hour post randomization between the 2 treatment arms separately for Group A and B
Platelet reactivity at 2 hours post randomization between the 2 treatment arms separately for Group A and B | 2 hours
  Platelet reactivity at 2 hours post randomization between the 2 treatment arms separately for Group A and B
Platelet reactivity at 4 hours post randomization between the 2 treatment arms separately for Group A and B | 4 hours
  Platelet reactivity at 4 hours post randomization between the 2 treatment arms separately for Group A and B
3. High on treatment platelet reactivity (HTPR) rates (≥208 PRU) at 0.5 hour post randomization between the 2 treatment arms, separately for Group A and B | 0.5 hour
  High on treatment platelet reactivity (HTPR) rates (≥208 PRU) at 0.5 hour post randomization between the 2 treatment arms, separately for Group A and B
High on treatment platelet reactivity (HTPR) rates (≥208 PRU) at 1 hour post randomization between the 2 treatment arms, separately for Group A and B | 1 hour
  High on treatment platelet reactivity (HTPR) rates (≥208 PRU) at 1 hour post randomization between the 2 treatment arms, separately for Group A and B
High on treatment platelet reactivity (HTPR) rates (≥208 PRU) at 2 hours post randomization between the 2 treatment arms, separately for Group A and B | 2 hours
  High on treatment platelet reactivity (HTPR) rates (≥208 PRU) at 2 hours post randomization between the 2 treatment arms, separately for Group A and B
High on treatment platelet reactivity (HTPR) rates (≥208 PRU) at 4 hours post randomization between the 2 treatment arms, separately for Group A and B | 4 hours
  High on treatment platelet reactivity (HTPR) rates (≥208 PRU) at 4 hours post randomization between the 2 treatment arms, separately for Group A and B
Occurrence of any 5-day bleeding event (BARC Types 1-5) | 5 days
  Occurrence of any 5-day bleeding event (BARC Types 1-5)
Occurrence of 5-day MACEs | 5 days
  Occurrence of 5-day MACEs

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Alexopoulos, MD, Principal Investigator — University Hospital of Patras
Locations (1):
- Cardiology Department Patras University Hospital, Rio, Achaia, Greece